CLINICAL TRIAL: NCT04199455
Title: The Differentiation and Treatment Scheme of TCM Key Syndromes for the Treatment of Acute Disabling Ischemic Stroke: a Randomized, Double-Blind, Placebo-Controlled Multicenter Trial
Brief Title: Evidence-based Evaluation of TCM Key Syndrome Differentiation and Treatment for Acute Ischemic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yefeng Cai, Director of Encephalopathy Center of Guangdong Provincial Hospital of Chinese Medcicine, Professor, Chief Physician, Neurologist, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018YFC1705002
Record Dates: First submitted 2019-12-08; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; neurologic impairment; integrative therapy; Chinese herbs; prospective randomized double-blind controlled trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Treatment Group (Experimental): Patients randomly assigned to the intervention group will receive EPACH and NQABC Chinese herbal compound granules, which will be manufactured by the Beijing Kangrentang Pharmaceutical company, combined with standard stroke care according to the Guidelines for the diagnosis and treatment of acute ischemic stroke in China 2018.
  Interventions: Drug: Integrative Treatment (EPACH Recipe Granules + NQABC Recipe Granules)
- Control Group (Placebo Comparator): Patients randomly assigned to the control group will receive recipe simulators as placebo, which will be manufactured by the Beijing Kangrentang Pharmaceutical company, combined with standard stroke care according to the Guidelines for the diagnosis and treatment of acute ischemic stroke in China 2018.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Integrative Treatment (EPACH Recipe Granules + NQABC Recipe Granules) — Patients randomly assigned to the intervention group will receive EPACH and NQABC Chinese herbal compound granules, which will be manufactured by the Beijing Kangrentang Pharmaceutical company, combined with standard stroke care according to the Guidelines for the diagnosis and treatment of acute ischemic stroke in China 2018.
  Route of administration: oral.
  Dose regimen:
  Day 1 to Day 5: in addition to the guideline-based standard treatment, 7.35g of EPACH recipe granules, dissolved with 200ml of boiled water, twice a day.
  Day 6 to Day 15: in addition to the guideline-based standard treatment, 6.85g of NQABC recipe granules, dissolved with 200ml of boiled water, twice a day.
  Other Names: EPACH Recipe Granules + NQABC Recipe Granules
  Arms: Integrative Treatment Group
Drug: Placebo — Patients randomly assigned to the intervention group will receive recipe simulators as placebo. EPACH and NQABC granules and recipe simulators are indistinguishable, identical in size, shape, color, appearance. Placebo is no decocting granules contain 5% original formula, 20% bitter gourd extract, 75% dextrin, and caramel color. Those who are assigned to the control group will be given placebo and guideline-based standard stroke treatment.
  Route of administration: oral.
  Dose regimen:
  Day 1 to Day 5: in addition to the guideline-based standard treatment, 7.35g of recipe simulator, dissolved with 200ml of boiled water, twice a day.
  Day 6 to Day 15: in addition to the guideline-based standard treatment, 6.85g of recipe simulator, dissolved with 200ml of boiled water, twice a day.
  Other Names: Recipe Simulators
  Arms: Control Group

SUMMARY:
The main purpose of this trial is to determine whether Chinese medicine (CM) for eliminating phlegm and clearing heat (EPACH) recipe continuously with nourishing Qi and activating blood circulation (NQABC) recipe, oral within 72 hours of symptom onset, improves the 15-day neurologicl deficits in participants with acute ischemic stroke.

DETAILED DESCRIPTION:
Many years of clinical practice experience has found that Chinese medicine (CM) for EPACH recipe continuously with NQABC recipe can be beneficial to the recovery of neurological function in the early stage of ischemic stroke. However, there is lack of high-quality evidence of its efficacy for acute ischemic stroke currently. The primary hypothesis of this trial is that Chinese herbal therapeutic regimen of EPACH+NQABC combined with guideline-based standard treatment will improve the 15-day neurological deficits in patients with acute ischemic stroke (AIS). Totally 500 participants will be randomized to the integrative treatment group treated with EPACH + NQABC recipes granules in addition to guideline-based standard treatment or the control group with placebo and guideline-based standard treatment equally for 15 days. All patients will have a National Institutes of Health Stroke Scale (NIHSS) entry score of 4-25. Patients in each group will be treated according to guideline-based standard treatment, but patients who have received or intend to undergo intravenous thrombolysis or endovascular interventions (including intravascular mechanical thrombectomy, arterial thrombolysis, angioplasty) are excluded. The primary outcome will be determined at 15 days, and all the participants will be followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Acute disabling ischemic stroke (4≤ NIHSS score ≤25 at the time of randomization) that can be treated with study drug within 72 hours of symptoms onset. Acute ischemic stroke, were confirmed by magnetic resonance imaging (MRI) or computer tomography (CT).
* Adult subjects (male or female ≥ 40 years and ≤ 80 years)
* Diagnosis of phlegm-dampness syndrome with manifestation of heat (the score of "Phlegm-dampness syndrome" ≥10 with the score of "Internal fire syndrome" ≥2 in Diagnostic Scale for Syndrome Elements of Ischemic Stroke.
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Planned or already receiving intravenous thrombolysis or endovascular treatment (intravascular mechanical thrombectomy, intra-arterial thrombolysis and angioplasty).
* Patients who have received other traditional Chinese Medicine Decoctions (Granules) and Chinese patent medicines Treatment for stroke.
* Confirmed secondary stroke caused by tumors, brain trauma, hematological diseases, infectious diseases, hereditary diseases, rheumatic immune diseases, etc
* modified Rankin Scale (mRS) Score > 2 at randomization (pre-morbid historical assessment).
* Other conditions that lead to motor dysfunction (i.n., severe osteoarthritis, rheumatoid arthritis, gouty arthritis, etc).
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) value that is twice the upper limit of normal)
* Severe non-cardiovascular comorbidity with life expectancy < 3 months.
* Complicated with other diseases that limited the evaluation of neurological function or affect the follow-up of patients.
* Known to be pregnant or breastfeeding.
* Currently receiving an investigational drug.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the change in the NIHSS scores from baseline to 15 days in the two groups. | Baseline and 15 days.
  The NIHSS score ranges from 0 (best score) to 42 (worst score).

SECONDARY OUTCOMES:
Proportion of Patients Independent | 30 days and 90 days after symptom onset.
  Proportion of patients independent is defined as Modified Rankin Scale score of 0, 1, or 2.
Activities of Daily Living | 30 days and 90 days after symptom onset.
  The Barthel Index score ranges from 0 (worst score) to 100 (best score).
Stoke Syndrome Factor Evaluation Scale | 5 days and 15 days after randomization.
  The Stroke Syndrome Factor Evaluation Scale ( a preliminary scale) is formed based on item response theory． It contains 76 items，among which there are 8 items of endogenous wind syndrome，24 items of endogenous fire syndrome, 12 items of phlegm-dampness syndrome, 8 items of blood stasis syndrome, 15 items of Qi deficiency syndrome, and 9 items of Yin deficiency syndrome．
Patient Reported Outcome (PRO) Scale of Stroke | 15 days after randomization
  PRO score ranges from 36 (best score) to 180 (worst score). PRO consists of four dimensions including the influence on physical, emotional, and social functioning, as well as the overall satisfaction with treatment.
Proportion of complications during hospitalization | During the period of hospitalization, an average of 10 to 15 days
  The complications include hemorrhagic transformation, pulmonary infection, urinary tract infection, Gastrointestinal hemorrhage, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yefeng Cai, MD, Principal Investigator — Guangzhou University of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No